CLINICAL TRIAL: NCT05209633
Title: Efficacy and Safety of Using Granules Dendrobii for the Treatment of Chronic Atrophic Gastritis in Subjects With Deficiency of Qi and Yin: a Randomized, Double-blind, Parallel, Placebo-controlled Study
Brief Title: Efficacy and Safety of Using Granules Dendrobii for the Treatment of Chronic Atrophic Gastritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Atrophic Gastritis Study
Record Dates: First submitted 2021-12-01; First posted 2022-01-26 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Atrophic Gastritis
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Granules Dendrobii) (Experimental): 6g each, 3 times per day, total 18 weeks
  Interventions: Drug: Granules Dendrobii
- Placebo (Placebo Comparator): 6g each, 3 times per day, total 18 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Granules Dendrobii — 6g each, 3 times per day, total 18 weeks
  Other Names: Dendrobii
  Arms: Active treatment (Granules Dendrobii)
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
Chronic atrophic gastritis (CAG) is a common and frequently-occurring disease, characterized by atrophy of gastric mucosal epithelium and glands, thinning of the mucosa, thickening of the submucosal muscle layer, intestinal metaplasia, and atypical hyperplasia. The course of the disease is protracted and often recurrent, which seriously affects the work and physical and mental health of the patient. Moreover, epidemiological studies have shown that the risk of gastric cancer in patients with chronic multifocal atrophic gastritis is significantly higher than that of the general population. Because CAG intestinal metaplasia and dysplasia can easily develop into gastric cancer, the World Health Organization (WHO) listed CAG's gastric mucosal atrophy, intestinal metaplasia and dysplasia as precancerous lesions of gastric cancer in 1978. Therefore, reversing and disappearing the precancerous state of gastric cancer is an effective measure to prevent the occurrence of gastric cancer.

The cause of CAG is complicated. Modern medicine believes that CAG is closely related to biological factors, physical and chemical factors, immune factors, and genetic factors. At present, there is no specific treatment, but symptomatic treatment is the main treatment. The disease belongs to the categories of "stomach pain" and "suffocation" in traditional Chinese medicine.

In many years of surveys and studies in Mainland China, it is found that Dendrobii granules have a good effect on chronic atrophic gastritis. It is planned to explore the possibility, effectiveness and safety of Dendrobii granules in the treatment of chronic atrophic gastritis through clinical trials.

20 subjects will be randomized into the treatment group and placebo group with 18 weeks of treatment.

DETAILED DESCRIPTION:
Chronic atrophic gastritis, (CAG) is a common and frequently-occurring disease, characterized by atrophy of gastric mucosal epithelium and glands, thinning of the mucosa, thickening of the submucosal muscle layer, intestinal metaplasia, and atypical hyperplasia. The course of the disease is protracted and often recurrent, which seriously affects the work and physical and mental health of the patient. Moreover, epidemiological studies have shown that the risk of gastric cancer in patients with chronic multifocal atrophic gastritis is significantly higher than that of the general population. Because CAG intestinal metaplasia and dysplasia can easily develop into gastric cancer, the World Health Organization (WHO) listed CAG's gastric mucosal atrophy, intestinal metaplasia and dysplasia as precancerous lesions of gastric cancer in 1978. Therefore, reversing and disappearing the precancerous state of gastric cancer is an effective measure to prevent the occurrence of gastric cancer. The study of CAG gastric mucosal atrophy and intestinal metaplasia reversal drugs not only has important academic significance, but also has good social and economic benefits, and has a broad market prospect.

The cause of CAG is complicated. Modern medicine believes that CAG is closely related to biological factors, physical and chemical factors, immune factors, and genetic factors. At present, there is no specific treatment, but symptomatic treatment is the main treatment. The disease belongs to the categories of "stomach pain" and "suffocation" in traditional Chinese medicine. The Chinese Medicine practitioners in the past have advocated that the main treatment is to nourish the stomach.

For more than two thousand years, a better understanding of Dendrobii used for "thick intestines and stomach", "calm the stomach", "replenish five internal organs and fatigue", and "light body and prolong life". There are many varieties of Dendrobii, especially Dendrobii officinale is the top grade. Dendrobii candidum is combined with American ginseng to nourish qi and nourish yin, nourish the stomach and promote fluid, nourish but not greasy, clear but not hurt the stomach.

This study used the Granules Dendrobii produced by Zhejiang Tianhuang Medical Plant Pharmaceutical Co., Ltd. (Hong Kong proprietary Chinese medicine registration number: HKC-16115). Granules Dendrobii has completed many pharmacodynamic and toxicological studies. In the many years of market investigation and research in Mainland China, it is found that Granules Dendrobii (Hong Kong Chinese Patent Medicine Registration Number: HKC-16115) has a good effect on chronic atrophic gastritis. Granules Dendrobii is suitable for the long-term conditioning and rehabilitation of spleen and stomach diseases that are weakened by spleen and stomach, or due to deficiency and solidification, resulting in spleen and stomach diseases mixed with deficiency and solid. Granules] with Dendrobium candidum as the main ingredient in the treatment of chronic atrophic gastritis has the traditional theoretical basis of Chinese medicine. Now plan to explore the possibility, effectiveness and safety of Granules Dendrobii in the treatment of chronic atrophic gastritis (qi and yin deficiency) through clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the diagnosis of chronic atrophic gastritis;
* TCM syndrome differentiation is deficiency of both qi and yin;
* Aged between 18 and 65 years old, regardless of gender;
* Volunteer to participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

* Patients with peptic ulcer, acid reflux, etc. who need PPI treatment;
* Patients with high-grade intraepithelial neoplasia of gastric mucosa or suspected malignant transformation in pathological diagnosis;
* Those who have received anti-HP treatment and related treatments in the past two weeks;
* Diabetic patients;
* Patients with severe heart, liver, kidney, lung, blood system diseases, abnormal renal function Cr test with clinical significance, and liver function ALT ≥ 1.5 times the upper limit of the normal reference value;
* People with allergies or a history of allergies to multiple drugs (two or more or the known ingredients in the drug);
* Those planning to become pregnant, pregnant or breast-feeding;
* Patients with mental illness;
* Those who have participated in other drug clinical trials within the past 3 months;
* The investigator believes that it is not suitable to participate in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change of histopathological grading of gastric mucosal atrophy. | 18 weeks
  Measure the improvement rate of histopathological grading of gastric mucosal atrophy.

SECONDARY OUTCOMES:
Histopathological changes of gastric mucosa | 18 weeks
  Other histopathological changes of gastric mucosa (intestinal metaplasia, dysplasia, chronic inflammatory reaction, activity, HP infection) grade changes by using the Visual Analogue Scale of New Sydney System. Mild, moderate and severe will be the grading of severity.
Grading changes of gastric mucosa | 18 weeks
  Changes in the grading of the gastric mucosa of gastric antrum (including gastric angle) and gastric body (atrophy, intestinal metaplasia, dysplasia, chronic inflammatory reaction, activity, HP infection) by using the Visual Analogue Scale of New Sydney System. Mild, moderate and severe will be the grading of severity.
Grading changes of epigastric bloating | 18 weeks
  The severity of epigastric bloating will be measured by using the scores 0,2,4,6. Which 0 means no symptom and 6 means most severe.
  Three gradings will be recorded: Symptom disappeared, improving or unchanged. Symptom disappeared means the score return to 0. Improving means the score decreases from baseline. Unchanged means score remain the same with baseline.
Grading changes of epigastric pain | 18 weeks
  The severity of epigastric pain will be measured by using the scores 0,2,4,6. Which 0 means no symptom and 6 means most severe.
  Three gradings will be recorded: Symptom disappeared, improving or unchanged. Symptom disappeared means the score return to 0. Improving means the score decreases from baseline. Unchanged means score remain the same with baseline.
The efficacy of TCM syndromes | 18 weeks
  Traditional Chinese Medicine syndromes such as epigastric bloating, epigastric pain, belching, loss of appetite will be assessed by the Chinese Medicine Practitioner. 4 gradings 0,1,2,3 will be used, which 3 is the most severe.
Inflammation changes under OGD | 18 weeks
  The severity of inflammation of gastric mucosa will be assessed under endoscopy. Four gradings of the severity which are normal, mild, moderate and severe according to the Visual Analogue Scale of New Sydney System.
The H. Pylori eradication rate | 18 weeks
  The H. Pylori eradication rate (positive at baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, Professor, Principal Investigator — Hong Kong Institute of Integrative Medicine
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No